CLINICAL TRIAL: NCT00435981
Title: A Phase II, Randomised, Double-Blind, Placebo-Controlled, Multi-Centre Study to Investigate the Impact of Diamyd® on the Progression of Diabetes in Patients Newly Diagnosed With Type 1 Diabetes Mellitus
Brief Title: Efficacy and Safety of Diamyd® in Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diamyd Therapeutics AB (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D/P2/04/3; EUDRACT 2004-003764-30
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; GAD65; Autoimmunity; C-peptide; Children
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases | interventions — Aluminum Hydroxide

INTERVENTIONS:
Drug: rhGAD65 formulated in Alhydrogel® (Diamyd®)

SUMMARY:
This is a randomized, placebo-controlled phase II study to investigate if a prime and boost of 20ug Diamyd® (rhGAD65 formulated in Alhydrogel®), administered subcutaneously four weeks apart, is safe and can preserve beta cell function in children and adolescents with type 1 diabetes with a diabetes duration less than 18 months at intervention.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients between 10 and 18 years of age, diagnosed with type 1 diabetes within 18 months
* Fasting C-peptide level above 0.1 nmol/l
* Presence of GAD65 antibodies
* Written informed consent (patient and parent/guardian)

Key Exclusion Criteria:

* Secondary diabetes mellitus or MODY
* Treatment with immunosuppressants
* Treatment with any vaccine within 1 month prior to first Diamyd® dose or planned treatment with vaccine up to 2 months after the second Diamyd® dose
* Participation in other clinical trials with a new chemical entity within the previous 3 months
* History of certain diseases or conditions (e.g. epilepsy, anaemia, alcohole or drug abuse)
* HIV or hepatitis
* Presence of associated serious disease or condition which in the opinion of the investigator makes the patient non-eligible for the study
* Pregnancy (or planned pregnancy within one year after 2nd administration)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70
Dates: Start 2005-01; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Diamyd® 20ug versus placebo with respect to preserving residual insulin secretion as measured by C-peptide levels. The effect of intervention will be evaluated at month 15 (main study period) and at month 30 (Extension phase).

SECONDARY OUTCOMES:
To evaluate the safety of Diamyd® 20ug.

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ludvigsson, MD, PhD, Principal Investigator — Div of Pediatrics, Dept of Clinical and Molecular Medicine, Faculty of Health Sciences, Linkoping University, Sweden
Locations (8):
- Sweden (8):
  - Borås Hospital, Borås
  - The Queen Silvia Children´s Hospital, Gothenburg
  - Halmstad Hospital, Halmstad
  - Ryhov Hospital, Jönköping
  - Linköping University, Linköping
  - University Hospital, MAS, Malmo
  - Örebro University Hospital, Örebro
  - Astrid Lindgren Children´s Hospital, Stockholm

REFERENCES:
- [Derived] Ludvigsson J, Cheramy M, Axelsson S, Pihl M, Akerman L, Casas R; Clinical GAD-Study Group in Sweden. GAD-treatment of children and adolescents with recent-onset type 1 diabetes preserves residual insulin secretion after 30 months. Diabetes Metab Res Rev. 2014 Jul;30(5):405-14. doi: 10.1002/dmrr.2503. PMID 24302596
- [Derived] Ludvigsson J, Hjorth M, Cheramy M, Axelsson S, Pihl M, Forsander G, Nilsson NO, Samuelsson BO, Wood T, Aman J, Ortqvist E, Casas R. Extended evaluation of the safety and efficacy of GAD treatment of children and adolescents with recent-onset type 1 diabetes: a randomised controlled trial. Diabetologia. 2011 Mar;54(3):634-40. doi: 10.1007/s00125-010-1988-1. Epub 2010 Nov 30. PMID 21116604
- [Derived] Ludvigsson J, Faresjo M, Hjorth M, Axelsson S, Cheramy M, Pihl M, Vaarala O, Forsander G, Ivarsson S, Johansson C, Lindh A, Nilsson NO, Aman J, Ortqvist E, Zerhouni P, Casas R. GAD treatment and insulin secretion in recent-onset type 1 diabetes. N Engl J Med. 2008 Oct 30;359(18):1909-20. doi: 10.1056/NEJMoa0804328. Epub 2008 Oct 8. PMID 18843118